CLINICAL TRIAL: NCT04216719
Title: Facilitating Opioid Care Connections: System Level Strategies to Improve Use of Medication-Assisted Treatment (MAT) and Movement Through the Opioid Care Cascade for Defendants in a New Opioid Court System
Brief Title: Facilitating Opioid Care Connections
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Center for Court Innovation (Other); New York State Unified Court System (Unknown); Center on Addiction (Unknown); Columbia University (Other); Weill Medical College of Cornell University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Katherine Elkington, Associate Professor of Clinical Medical Psychology, in Psychiatry, Co-Director, Center for the Promotion of Mental Health in Juvenile Justice, Division of Child and Adolescent Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 7872; UG1DA050071 (NIH)
Record Dates: First submitted 2019-12-19; First posted 2020-01-03 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Opioid Court Model; Medication to Treat Opioid Use Disorder; Opioid Use

STUDY DESIGN:
Intervention Model Description: Stepped-wedge design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OCM-RISE (Experimental): Opioid court team provided external facilitation to generate action plans to develop and roll out or improve practice of the county opioid court.
  Interventions: Behavioral: OCM-RISE

INTERVENTIONS:
Behavioral: OCM-RISE — OCM RISE will comprise four phases (Exploratory, Preparation, Implementation, and Sustainment). During Exploration, staff will conduct readiness surveys, interviews and system mapping exercises to assess county context. In the Preparation Phase, the needs assessment data will inform county-specific action plans. Guided facilitation during this phase includes court development planning, practice/process improvement strategies, and training on data-driven decision-making to help IACTs operationalize the 10 OCM guidelines, assess performance, and fit the guideline to the local context. In the Implementation Phase, counties will roll out the OCM for 18 months with data feedback, support, and facilitation. Each IACT will receive reports on the performance of its OCM and complete two plan-do-study-act cycles. In the Sustainment Phase, implementation and feedback reports will continue for 6-18 months, but without other external facilitation.

SUMMARY:
In response to the opioid crisis in New York State (NYS), where the propose project will take place, the Unified Court System (UCS) developed a new treatment court model - the opioid court model (OCM) - designed around 10 practice guidelines to address the flaws of existing drug courts and reduce overdose (OD), opioid use disorder (OUD), and recidivism via rapid screening and linkage to medication for opioid use disorder (MOUD). In 2018, NYS began to expand the OCM across NYS. Yet, given the innovation of the OCM, the exact barriers to implementation in disparate counties with a range of resources - and the strategies to overcome them - are largely unknown. The research team proposes to integrate evidence-based implementation strategies to refine and evaluate the Opioid Court Model Rigorous Implementation Science for Effectiveness (OCM RISE) intervention, an implementation intervention that will allow the OCM, as framed by the 10 practice guidelines, to be scaled up across NYS.

DETAILED DESCRIPTION:
Aims. Guided by Exploration Preparation Implementation Sustainment (EPIS) model and Social Cognitive Theory (SCT), Specific Aims are: 1) To refine OCM-RISE using mixed-method formative work with 5 NYS "initial adopter" counties, who established opioid courts before 2019, that (a) identifies gaps in service provision by documenting OCM/opioid cascade outcomes; (b) identifies successes/challenges in operationalizing guidelines; and (c) characterizes the working relationships between county opioid court and treatment systems. 2). In a cluster-randomized, stepped-wedge design in 10 "new adopter" counties, which includes some counties who established opioid courts in 2019, compared to baseline treatment as usual (drug courts), test, (a) the implementation impact of OCM RISE in improving implementation outcomes along the opioid cascade (screening/identification, referral, treatment enrollment, MOUD initiation); and (b) the clinical and cost effectiveness of OCM RISE in improving public health (treatment retention/court graduation) and public safety (recidivism) outcomes, exploring moderators: defendant gender, age, charge; county urbanicity and county OD rates. 3) To characterize and compare advancement through the stages of implementation of the OCM in the 10 counties, elucidating the inner- and outer-level EPIS- and SCT-derived factors that influence delivery of implementation strategies to inform OCM scale up; and (b) to explore the relationship between implementation stage completion and all opioid cascade, public health and public safety outcomes.

Setting.The research team will leverage the real-world roll-out of the OCM by the NYS UCS to provide implementation strategies that will optimize the ability of diverse counties to effectively adopt this innovative model. Between 2017 and 2019, several counties have scaled up these courts, and the research team will use their experiences and outcomes in intervention refinement. The team will then evaluate OCM RISE in 10 "new adopter" counties, some if which have established opioid courts in 2019, that all have an existing adult drug (non-opioid) court. Counties are varied in their experience of opioid "burden" as well as the stage of the development of their court.

Design, Sample Size and Randomization. In the proposed cluster randomized stepped-wedge design, 10 new adopter counties will be randomized - stratified by population density/urbanicity (as a proxy for staffing and resource availability), (a metric developed by NYS Department of Health (DOH) that encompasses non-fatal ER visits and hospital discharges involving opioid use, OD deaths, which will be used as a proxy for treatment need), and county court activity (newly established versus not)- to one of 5 waves of OCM RISE at 2-month intervals. The 2-month intervals for randomization reflect the real world need for counties to meet the UCS mandate to establish opioid courts as well as our experience with managing multiple start-ups across NYS. The research team will examine the differences between matched defendants with opioid use (OU) or OUD at baseline (county drug court outcomes in the 3 months prior to randomization) with those after OCM RISE on opioid cascade outcomes and on recidivism. By randomizing sites across time, the control group is taken to be counties that have not yet been randomized by a particular time, i.e., treatment as usual (TAU), allowing us to control for secular changes over time. During the pre-randomization period the opioid cascade outcomes will be collected on defendants with OU or OUD who enter into the existing county drug courts. The team expects that introduction of the OCM will identify a broader case-mix of defendants with OU than those currently identified for drug courts.

Hence, the research team will take into account defendant level differences (e.g. heroin vs prescription drug use, age, OUD severity) when testing the effect of OCM by using propensity score matching. There are two limitations to cluster randomized deigns: potential of uneven distribution of potentially confounding variables within a cluster (i.e. county) as well as interrelationship between variables. Our proposed stratification plan and use of propensity matching will address issues related to confounding. The team calculated our ability to detect an effect of the OCM (i.e. power) using a conservative intraclass correlation coefficient (ICC) of 0.05 denoting a moderate positive correlation between outcomes within a county to address issues of interrelationship between variables at the county level

Participants. Participants will be court and treatment staff who participate in 1) staff surveys, 2) in-depth interviews, 3) focus groups, 4) the interagency change team (IACT) and/or 5) preparation activities (e.g. leadership meeting, orientation meeting). Approximately n=10 court and n=10 treatment staff will be recruited in each county for a total of 200 participants. Main study outcome data are to be drawn from court records of defendants, who are not considered human subjects and will not be enrolled in the study.

Formative Phase (with "initial adopter" counties). Convene expert stakeholder OCM Advisory Panel with "initial adopter" counties. At the outset of the grant, the team will convene an OCM Advisory Panel of stakeholders involved in OCM implementation in 5 counties who implemented opioid courts before 2019. In a half-day meeting at each county, the research team will lead discussion of facilitators and barriers relevant to each step of the opioid care cascade. Stakeholders will discuss experiences, facilitators, and barriers in operationalizing the UCS OCM practice guidelines (and meeting benchmarks if set) in their counties. This discussion will inform development of a set of benchmarks for the 10 OCM RISE guidelines. These data will contribute to identifying specific areas of focus for the proposed implementation intervention (OCM RISE) and informing needed changes or refinements.

Intervention Phases (with "new adopter" counties). OCM RISE will comprise four phases (Exploratory, Preparation, Implementation, and Sustainment) that a new adopter county will use to roll out the OCM. OCM RISE implementation strategies, grouped to achieve three implementation goals, have been well documented in projects that involve interagency collaboration and/or delivery of evidence-based guidelines, and use of data to guide decision- making and improve current practices has been successfully implemented in justice (e.g., JJTRIALS), health, education, and business settings. In the Exploratory Phase (5 months), research staff will conduct readiness surveys, system mapping exercises, focus groups and in-depth interviews to assess county context to allow specific content of implementation strategies to be tailored to that county's needs and capabilities. The research team will integrate these data to prepare a needs assessment report to be presented to each county's court and treatment leadership in the Preparation Phase (7 months) and be used by the Inter Agency Change Team (IACT), with guidance from external facilitators, to create an implementation plan for the county. Guided facilitation during this phase will include court development planning for counties without opioid courts and practice and process improvement planning to help all IACTs operationalize the 10 OCM guidelines and achieve a balance between fidelity to the guideline and fit to the local context; and training on data-driven decision-making (DDDM) to allow IACTs to use data to inform continued process improvement and practice changes to optimize OCM delivery. DDDM is a process, frequently used in the justice system, by which key system stakeholders collect, analyze, and interpret data to inform decisions that will help improve a range of outcomes/practices. In the Implementation Phase (18 months), the county will roll out the OCM for 18 months with data feedback, support, and facilitation from the research team. Each IACT will be provided with data on performance of its county OCM following implementation, and complete two plan-do-study-act (PDSA) cycles. PDSA is an evidence-based, rapid-cycle change model for testing organizational enhancements on a small scale before incorporating them on a larger scale. It is a flexible modality that can be used to achieve sustainable quality improvement and may be particularly useful in a court system that requires evidence before policy or procedures are altered. In the Sustainment Phase (6-18 months depending on the study wave), OCM implementation and feedback reports will continue but without other external facilitation.

Assessments and analysis. Data sources in the proposed study include court system records (Unified Case Management System; UCMS), staff surveys, focus groups and checklists. Staff surveys are administered at 3 timepoints: during baseline data collection (before exploration or preparation being), at the beginning of the implementation phase and at the end of the sustainment phase. Main outcome data will be drawn from the UCMS. The research team will determine the clinical effectiveness of OCM RISE by determining differences between matched defendants with OU or OUD in county drug courts (baseline) with those in the OCM on (i) retention in community treatment for >60 days/court completion (primary outcome) and recidivism 6 months after OCM termination/graduation; cost- effectiveness will also examine abstinence. The research team will examine the implementation impact of OCM RISE by examining differences between matched defendants with OU or OUD in county drug courts (baseline) with those in the OCM on (i) identification of service need; (ii) referral to community-based treatment/MOUD; (iii) enrollment in treatment/MOUD; (iv) MOUD initiation. By randomizing sites to OCM-RISE across time, the control group (which is changing over time) is taken to be the sites that have not yet rolled out the OCM by a particular time, treatment as usual (TAU).

Clinical effectiveness and Implementation impact will be determined using generalized linear mixed effects modeling for stepped-wedge designs. In the event that descriptive analyses identify large differences in the case mix of background characteristics for the defendants during the TAU period prior to OCM implementation as compared to the case-mix after OCM implementation, the team will additionally implement propensity score matching. Cost effectiveness will be determined using multivariable Generalized Linear Mixed Model. The multivariable aspect of the model allows for the control of potentially confounding factors that are unbalanced between arms because they either were not accounted for in the randomization process or became unbalanced due to loss to follow-up. EPIS and SCT derived inner and outer setting factors will be examined as mediators and moderators in clinical effectiveness and implementation impact analysis; data are derived from staff surveys.

To explore the implementation process, the team will characterize the paths through stages of implementation through to sustainability, as measured by the Stages of Implementation Change (SIC) tool, across counties, exploring differences between counties that have recently implemented a new opioid court (within 2019) prior to study participation and counties that had not. Through case studies the team will qualitatively describe how different counties deal with the different barriers they face and progress through the implementation phases. The research team will combine quantitative and qualitative data collected throughout the implementation process from multiple sources, including: in-depth interviews, UCMS data, staff surveys, and county data.

ELIGIBILITY:
Court Staff

Inclusion Criteria:

* Employed by the Unified Court System/County Court in participating county
* Age 18+
* Understands and speaks English

Exclusion Criteria:

- None

County Treatment Staff Inclusion Criteria

* Employed at substance use (SU) treatment agency
* Age 18+
* Understands and speaks English

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3440 (Estimated)
Dates: Start 2020-03-18 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who are retained in treatment for at least 60 days | Through study completion, an average of 30 months
  Derived from Unified Court Management System (UCMS)
Number of participants who graduate from court | Through study completion, an average of 30 months
  Derived from Unified Court Management System (UCMS)
Number of participants who are abstinent from opioid use | Through study completion, an average of 30 months
  Derived from Unified Court Management System (UCMS)
Number of participants who recidivate within 12 months following court completion | Through study completion, an average of 30 months
  Derived from Unified Court Management System (UCMS)

SECONDARY OUTCOMES:
Number of defendants who are screened for opioid use after arrest | Through study completion, an average of 30 months
  Derived from Unified Court Management System (UCMS)
Number of court participants who are referred for opioid treatment | Through study completion, an average of 30 months
  Unified Court System Management Information System (UCMS)
Number of court participants who are provided medication for Opioid Use Disorder (MOUD) Initiation | Through study completion, an average of 30 months
  Unified Court System Management Information System; UCMS data field
Acceptability of the opioid court | At study completion
  Opinions of acceptability of OCM RISE as derived from a focus group with interagency change team members
Adoption of OCM RISE | Through study completion, an average of 30 months
  Number of implementation stages (as determined by EPIS: exploration, preparation, implementation, sustainment) completed measured by the Stages if Implementation Completion (SIC) tool
Sustainability of OCM RISE | Through study completion, an average of 30 months
  Continued screening, referral, treatment enrollment, MOUD initiation 12m post Implementation phase ends

OTHER OUTCOMES:
Knowledge, Attitudes towards MOUD | Through study completion, an average of 30 months
  Court and Treatment Staff Survey
Self-Efficacy to address Opioid Use Disorder | Through study completion, an average of 30 months
  Court and Treatment Staff Survey
Perceived Importance of Cascade Behaviors | Through study completion, an average of 30 months
  Court and Treatment Staff Survey
Perceived Potential Sustainability of OCM | Through study completion, an average of 30 months
  Court and Treatment Staff Survey
Practice change | Through study completion, an average of 30 months
  Training quiz
Organizational climate, support, and functioning | Through study completion, an average of 30 months
  Court and Treatment Staff Survey
Leadership innovation | Through study completion, an average of 30 months
  Court and Treatment Staff Survey
Inter-agency Organizational Features | Through study completion, an average of 30 months
  Court and Treatment Staff Survey
Structural Organizational Characteristics | Through study completion, an average of 30 months
  Bi-Monthly check-ins; Readiness Survey
Defendant Characteristics | Through study completion, an average of 30 months
  Unified Court System Management Information System; UCMS data field;

CONTACTS AND LOCATIONS:
Overall Officials: Katherine S Elkington, PhD, Principal Investigator — Columbia University/NYSPI; Edward Nunes, MD, Principal Investigator — Columbia University/NYSPI; Milton L Wainberg, MD, Principal Investigator — Columbia University/NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States